CLINICAL TRIAL: NCT02374229
Title: Surgical Ablation of Ganglion Plexuses of the Pulmonary Artery in Patients With Valvular Heart Disease, Complicated by High Pulmonary Hypertension May Reduce Its Degree.
Brief Title: Ablation of the Pulmonary Artery With High Pulmonary Hypertension During Mitral Valve Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAPA 1
Record Dates: First submitted 2015-02-12; First posted 2015-02-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; pulmonary artery denervation; mitral valve disease
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Radiofrequency Ablation; Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The study group (Experimental): Procedure: mitral valve surgery, surgical ablation of ganglion plexus pulmonary artery.
  Will include 15 patients with mitral stenosis or insufficiency subject to correction, complicated by high pulmonary hypertension. During the operation, a standard surgical procedure for the treatment of heart valve disease will be complemented by the ablation zone of bifurcation of the pulmonary artery, surgical ablation of ganglion plexus pulmonary artery.
  For mitral regurgitation or stenosis, the procedures will be a valve repair or mitral valve replacement.
  Procedure will be considered effective in the face of declining average pressure in the pulmonary artery for invasive monitoring of 10mm Hg and more.
  Interventions: Procedure: Surgical ablation of ganglion plexus pulmonary artery.; Procedure: mitral valve surgery
- The control group (Active Comparator): Procedure:mitral valve surgery. Will include 15 patients with mitral stenosis or insufficiency subject to correction, complicated by high pulmonary hypertension. Patients will be made standard procedure correction mitral valve disease without pulmonary artery denervation.
  For mitral regurgitation or stenosis, the procedures will be a valve repair or mitral valve replacement only.
  Interventions: Procedure: mitral valve surgery

INTERVENTIONS:
Procedure: Surgical ablation of ganglion plexus pulmonary artery. — Performed ablation zone pulmonary artery bifurcation, at 2mm proximal direction and a distal direction in the left and right branches of the pulmonary artery using the electrophysiological device Atricure.
  Other Names: surgical ablation; radiofrequency ablation
  Arms: The study group
Procedure: mitral valve surgery — The standard procedure for mitral regurgitation or stenosis, the procedures will be a valve repair or mitral valve replacement, depending upon the particular morphological condition of the mitral valve.
  Other Names: mitral valve repair; mitral velve replacement

SUMMARY:
The aim of this prospective randomized study was to evaluate the effectiveness and safety of the original ablation procedures ganglion plexus pulmonary artery with simultaneous correction of valvular heart disease, complicated by high pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension is a serious condition, the severity of which is often underestimated. About 10% of significant mitral heart disease complicated by high pulmonary hypertension (more than 60 mm Hg). Up to 70% of patients retain this level of pulmonary hypertension after successful treatment of heart valve disease.The quality of life of patients with persistent high pulmonary hypertension is significantly lower than in patients with mild to moderate degree. Risks of recurrent tricuspid insufficiency and right ventricular dysfunction is much higher. Despite the use of modern drug therapy of pulmonary hypertension in patients with valvular heart disease satisfactory clinical effect is achieved only in a small number of patients. Our team proposed a new original method of ablation of the pulmonary artery with simultaneous open cardiac surgery correction of mitral heart disease in patients with high baseline pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mitral stenosis or insufficiency complicated by high pulmonary hypertension (mean pulmonary artery pressure in invasive monitoring more than 35 mm Hg), which are subject to surgical treatment.

Exclusion Criteria:

* pulmonary stenosis;
* pulmonary embolism in history;
* congenital heart disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Death of the patient | 3 weeks

SECONDARY OUTCOMES:
Mean pulmonary artery pressure in invasive monitoring | 3weeks; 6 and 12 months after the procedure.
  Patients will be installed catheter Swan-Ganz in the intensive care unit for invasive measurement of pulmonary artery pressure.
Exercise tolerance (the 6 minute walk test (6MWD) | 3weeks; 6 and 12 months after the procedure.
  the 6 minute walk test (6MWD)
quality of life | 3weeks; 6 and 12 months after the procedure.
  SF-36 questionnaire
adverse events | 3 weeks
  complications associated with the procedure plexus ganglion ablation, such as perforation of the pulmonary artery, pulmonary artery dissection, pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Bogachev-Prokophiev, MD PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Novosibirsk Oblast, Russia